CLINICAL TRIAL: NCT01177514
Title: The Role of Gabapentin in Postoperative Pain and Epithelialization After Photorefractive Keratectomy A Prospective, Randomized, Double Blinded, Placebo Controlled Study
Brief Title: The Role of Gabapentin in Postoperative Pain and Epithelialization After Photorefractive Keratectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Codet Vision Institute (Other)
Responsible Party: Principal Investigator, ALEJANDRO LICHTINGER, MD, Codet Vision Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GABA1
Record Dates: First submitted 2010-04-23; First posted 2010-08-09 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Pain After Photorefractive Keratectomy
Keywords: Refractive surgery; PRK; PAIN; Gabapentin
MeSH Terms: conditions — Pain | interventions — Gabapentin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GABAPENTIN (Experimental): Group of patients treated with oral gabapentin
  Interventions: Drug: Gabapentin
- PLACEBO (Placebo Comparator): Group given the placebo capsules
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Gabapentin — Gabapentin PO. (300MG) 1 capsule the night before surgery, q12hrs the day of surgery and q8hrs for the firt 3 postoperative days.
  Arms: GABAPENTIN
Drug: Sugar pill — Sugar pill. One capsule given the night before surgery, q12hrs on the day of surgery and q8hrs for the first 3 postoperative days.
  Arms: PLACEBO

SUMMARY:
The primary aims of this study are to determine if treatment with Gabapentin taken systemically (oral tablets) in patients who have photorefractive keratectomy (PRK) surgical treatments reduces post surgical neuropathic pain and discomfort. The investigators main Hypothesis is that gabapentin given prior to and after refractive surgery prevents central sensitization and local allodynia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age
2. Subjects must not have any corneal disease or degeneration
3. Subjects must be candidates for LASIK or PRK refractive surgery

Exclusion Criteria:

1. History of topical ocular medications within 4 weeks prior to enrollment
2. History of conjunctivitis or ocular inflammation within 4 weeks prior to enrollment
3. History of a previous refractive surgery
4. History of previous diagnosis of corneal disease, degeneration, or glaucoma
5. History of autoimmune disease
6. History of oral anti-histamines currently or within 1 week of study enrollment
7. History of systemic anti-inflammatory or pain medication currently or within 4 weeks of study enrollment
8. Use of oral diuretics or betablocker currently or within 1 week of study enrollment
9. Current diagnosis of dry eye
10. Patients whose Best corrected vision is less than 20/20
11. Patients whose target post operative refraction is not plano
12. Pregnant and lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pain at moment of examination | 24 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Average pain for the previous 24 hour period, | assesed at 24 hours
  Numerical visual scale questionnaire, a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
Maximum pain intensity for the previous 24 hour period | Assesed at 24 hours postoperatively
  In a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded.
Pain at moment of examination | 48 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
pain on examination | 72 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
pain on examination | 96 hours ostoiperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Pain at moment of examination | postoperative day 7
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Average pain for the previous 24 hour period | Assesed at 48 hours
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Average pain during the previous 24 hour period | Assesed at 72 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Average pain for the last 24 hours period | Assesed at 96 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Average pain since last examination | Assesed on postopertive day 7
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Maximum pain intensity for the previous 24 hour period | Assesed at 48 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Maximum pain intensity for the previous 24 hour period | Assesed at 72 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Maximum pain intensity for the last 24 hour period | Assesed at 96 hours postoperatively
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day
Maximum pain intensity since the last examination | Assesed on the 7th postoperative day
  Numerical Visual scale questionnaire. a scale from 0-10 where 0 is the least amount of pain and 10 being the most pain felt was recorded
  Every patient will be examined every 24 hours until complete healling which usualy takes place between 3 and 4 days; after complete healing the next and last examination is performed at the 7th postoperative day

SECONDARY OUTCOMES:
Time required for complete healing | Evaluated each day until complete healing
  Slit lamp observation of the epithelial defect and time until removal of contact lens.
Visual acuity | every day until complete healing and at the 7th day postop
  Snellen Chart
Foreign body sensation | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale, In a scale from 0-10 where 0 is the least amount of foreign body sensation and 10 being the most.
Light sensitivity | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale, in a scale from 0-10 where 0 is the least amount of light sensitibity and 10 being the most.
Tearing and watery eyes | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale questionaire, In a scale from 0-10 where 0 is the least amount of tearing and 10 being the most.
Eye discomfort | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale questionnaire, In a scale from 0-10 where 0 is the least amount of discomfort and 10 being the most.
Dizziness | Every 24 hours until complete healling and at the 7th day postop
  Numerical visual scale, scale from 0-10 where 0 is the least dizzy and 10 being the most.
lethargy | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale, In a scale from 0-10 where 0 is the least lethargic and 10 is the most.
Headache | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale, In a scale from 0-10 where 0 is the least amount of headache and 10 being the most severe headache felt.
Gastro-intestinal symptoms | Every 24 hours until complete healing and at the 7th day postop
  Numerical visual scale, In a scale from 0-10 where 0 is the least amount of symptoms and 10 being the most symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Codet Vision Institute, Tijuana, Estado de Baja California, Mexico